CLINICAL TRIAL: NCT03165617
Title: A Phase III/IV, Stratified, Randomized, Observer Blind, Multicenter Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of a Cell-Based Quadrivalent Subunit Influenza Virus Vaccine Compared to Non-Influenza Comparator Vaccine in Subjects ≥2 to <18 Years of Age
Brief Title: Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of QIVc in Subjects ≥2 to <18 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V130_12; 2016-002883-15 (EudraCT Number)
Record Dates: First submitted 2017-05-17; First posted 2017-05-24 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Influenza, Human
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Phase 3/4
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QIVc (≥2 years to <18 Years of Age) (Experimental): Cell-derived Seasonal Quadrivalent Influenza Vaccine
  Interventions: Biological: QIVc
- Non-Influenza Comparator Vaccine (Active Comparator): Non-Influenza Comparator Vaccine
  Interventions: Biological: Non-influenza Comparator Vaccine

INTERVENTIONS:
Biological: QIVc — Cell-derived Quadrivalent Influenza Vaccine for intramuscular use containing each of the 2 influenza type A strains and each of the 2 influenza type B strains
  Other Names: Flucelvax Quadrivalent
  Arms: QIVc (≥2 years to <18 Years of Age)
Biological: Non-influenza Comparator Vaccine — Non-influenza comparator vaccine for intramuscular use
  Arms: Non-Influenza Comparator Vaccine

SUMMARY:
This Phase 3/4, randomized, observer-blind, multi-center study, stratified study evaluated the immune (antibody) response, efficacy and safety of a cell-derived quadrivalent subunit influenza virus vaccine (Seqirus QIVc) in comparison with a non-influenza comparator, meningococcal serogroup A, C, W-135, and Y (Menveo®, GlaxoSmithKline Biologicals, S.A.) in healthy pediatric subjects ≥2 Years to <18 Years of Age

DETAILED DESCRIPTION:
This Phase 3/4, randomized, observer-blind, multi-center, stratified study evaluated the efficacy, safety, and immunogenicity of a cell-derived quadrivalent subunit influenza virus vaccine (Seqirus QIVc) compared to a non-influenza comparator vaccine in healthy male and female participants between 2 to <18 years of age. A total of 4514 children/teens were randomized, receiving either QIVc or the non-influenza comparator vaccine. The comparator was (meningococcal [Groups A, C, W-135, and Y] oligosaccharide diphtheria CRM197 conjugate vaccine [Men ACWY]). Randomized enrollment was stratified in a 1:1 ratio via an Interactive Response Technology (IRT) system which assigned the participants into two age cohorts: 2 to <9 years of age and 9 to <18 years of age. Subjects between 2 to <9 years of age were further stratified by previous influenza vaccine status ("previously vaccinated" or "not previously vaccinated").

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥2 to <18 years of age on the day of the first study vaccination
* Subject's parent(s) or legal guardian(s) who was/were able to give informed consent/dissent after the nature of the study had been explained in accordance with the practices described in the study and according to local regulatory requirements
* If the subject was of an age where, according to local regulations, informed assent was required, he/she must have provided assent to participate in the study
* Subject/subject's parent(s) or legal guardian(s) was/were able to comply with study procedures and was/were available for follow-up; and
* Subject was in generally good health as per the investigator's medical judgment

Exclusion Criteria:

* Clinical signs of fever and/or an oral temperature of ≥100.4°F (38.0°C) within 3 days prior to vaccination;
* A known history of any anaphylaxis, serious vaccine reactions or hypersensitivity to any of the vaccine components described in the Investigator's Brochure, or had any of the contraindications listed in the package insert of the comparator vaccine;
* A history of Guillain-Barré syndrome or other de-myelinating diseases such as encephalomyelitis and transverse myelitis;
* Female subject of childbearing potential (ie, post onset of menarche and before natural or induced menopause), sexually active, and who did not use any acceptable contraceptive methods for at least 2 months prior to study entry and who did not intend to use any acceptable contraceptive methods throughout subject participation (acceptable contraceptive methods included: abstinence; hormonal contraceptive [such as oral, injection, transdermal patch, implant]; diaphragm with spermicide; tubal occlusion device; intrauterine device [IUD]; tubal ligation; male partner using condom; or male partner having been vasectomized);
* Pregnant or breast feeding female;
* Subject and/or subject's parent/guardians who were not able to comprehend or follow all required study procedures for the entire period of the study;
* Received prior Meningococcal ACWY vaccination that conflicted with national recommendations or local practices for the timing of the primary or the booster vaccination;
* Received influenza vaccination or had documented influenza disease in the last 6 months;
* Known or suspected congenital or acquired immunodeficiency; or received immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or systemic corticosteroid therapy (prednisone or equivalent) at any dose for more than 2 consecutive weeks (14 days) within the past 3 months. Topical, inhaled and intra-nasal corticosteroids were permitted. Intermittent use (1 dose in 30 days) of intra-articular corticosteroids was also permitted;
* Administration of immunoglobulin and/or any blood products within the 3 months preceding vaccination, or administration was planned during the study;
* Participated in any clinical study with another investigational product within 30 days prior to first study visit or intended to participate in another clinical study at any time during the conduct of this study. Concomitant participation in an observational study (not involving drugs, vaccines, or medical devices) was acceptable;
* Medical conditions or treatments contraindicating IM vaccination due to increased risk of bleeding. These included known bleeding disorders (such as thrombocytopenia), or treatment with anticoagulants (such as warfarin) in the 3 weeks preceding vaccination. Antiplatelet agents such as low-dose aspirin, ticlopidine (Ticlid) and clopidogrel (Plavix) were permitted;
* Evidence or history (within the previous 12 months) of drug or alcohol abuse;
* Study personnel or immediate family members (brother, sister, child, parent), the spouse of study personnel or individuals who were financially or emotionally dependent on study staff;
* Participated in this study in a prior season, if applicable; or
* Any clinical condition that, in the opinion of the investigator, may have interfered with the results of the study or pose additional risk to the subject due to participation in the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4514 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (40):
- Australia (2):
  - 302 AusTrials Pty Ltd, Sherwood, Queensland
  - 300 Murdoch Childrens Research Institute, Carlton, Victoria
- Estonia (6):
  - 500 Merelahe Family Doctors Centre, Tallinn, Harju
  - 504 Merekivi Family Doctors Ltd, Tallinn, Harju
  - 502 Medicum AS, Tallinn, Harju
  - 503 Vee Family Doctors Centre, Paide, Järvamaa
  - 505 Clinical Research Center, Tartu, Tartu
  - 505 Clinical Research Center, Tartu
- Finland (10):
  - 607 Espoo Vaccine Research Clinic, Espoo
  - 603 Helsinki South Vaccine Research Clinic, Helsinki
  - 604 Helsinki South Vaccine Research Clinic, Helsinki
  - 600 Järvenpää Vaccine Research Clinic, Jarvenpaa
  - 606 Kokkola Vaccine Research Clinic, Kokkola
  - 605 Oulu Vaccine Research Clinic, Oulu
  - 601 Pori Vaccine Research Clinic, Pori
  - 602 Seinäjoki Vaccine Research Clinic, Seinäjoki
  - 608 Tampere Vaccine Research Clinic, Tampere
  - 609 Turku Vaccine Research Clinic, Turku
- Lithuania (6):
  - 706 Private Office of Children Pulmonologist, Alytus, Alytus Apskritis
  - 704 Kauno klinikine ligonine, Kaunas, Kaunas County
  - 703 UAB InMedica, Kaunas, Kaunas County
  - 702 JSC Saules seimos medicinos centras, Kaunas, Kaunas County
  - 700 Kaunas Silainiai Outpatient Clinic, Kaunas, Kauno Apskrits
  - 701 Naujininkai Outpatient Clinic, Vilnius, Vilnaius Apskritis
- Philippines (7):
  - 402 De La Salle Health Sciences Institute, Dasmariñas, Cavite
  - 405 De La Salle Health Sciences Institute, Dasmariñas, Cavite
  - 403 Philippine General Hospital, Manila, National Capital Region
  - 404 Philippine General Hospital, Manila, National Capital Region
  - 400 Research Institute For Tropical Medicine, Muntinlupa, National Capital Region
  - 401 Research Institute For Tropical Medicine, Muntinlupa, National Capital Region
  - 406 Research Institute For Tropical Medicine, Muntinlupa, National Capital Region
- Poland (6):
  - 805 Szpital Uniwersytecki nr 2 im. dr. Jana Biziela w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - 806 Specjalistyczny Szpital im. E. Szczeklika w Tarnowie, Tarnów, Lesser Poland Voivodeship
  - 803 Szpital im. Sw. Jadwigi Slaskiej w Trzebnicy, Trzebnica, Lower Silesian Voivodeship
  - 800 Niepubliczny Zaklad Opieki Zdrowotnej (NZOZ) "Salmed" s. c., Łęczna, Lublin Voivodeship
  - 804 Prywatny Gabinet Lekarski, Dębica, Podkarpackie Voivodeship
  - NZLA Michalkowice - Jarosz i Partnerzy Spolka Lekarska, Siemianowice Śląskie, Silesian Voivodeship
- 900 Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña, Spain
- Thailand (2):
  - 200 Srinagarind Hospital, Khon Kaen University, Khon Kaen, Muang
  - 201 ChiangMai University, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Seqirus supports the release of anonymized subject-level and study-level data in compliance with regulatory requirements, including Clinical Documents which are part of the CTD modules submitted to regulatory agencies for public release.
  Summary results disclosure is either in document form (e.g., ICH E3 Clinical Study Report synopsis) or structured data form (such as summary results in ClinicalTrials.gov (United States) or eudract.ema.europa.eu (EU Clinical Trial Registry [EU CTR]).
Supporting Information: Study Protocol, SAP
Time Frame: Seqirus aims to disclose these results from clinical studies within twelve (12) months of the Study Completion unless otherwise mandated by local law or regulation.
Access Criteria: All requests will be fully vetted and data to be released approved, prior to distribution. Seqirus does not release subject-level data and study-level data if the requester's purpose is to conduct a re-analysis of the study data, as opposed to a meta-analysis.
  While the URL link below does not outline the data sharing policy per se, it does present a high-level view of how the organization partners with external collaborators
URL: https://www.seqirus.com/partnering

REFERENCES:
- [Derived] Nolan T, Fortanier AC, Leav B, Poder A, Bravo LC, Szymanski HT, Heeringa M, Vermeulen W, Matassa V, Smolenov I, Edelman JM. Efficacy of a Cell-Culture-Derived Quadrivalent Influenza Vaccine in Children. N Engl J Med. 2021 Oct 14;385(16):1485-1495. doi: 10.1056/NEJMoa2024848. PMID 34644472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled over 3 seasons, starting in SH 2017, followed by NH 2017-2018 and NH 2018-2019. Recruitment was conducted in 8 countries over these 3 seasons: Australia, Philippines and Thailand (Season 1); Estonia and Finland i(Season 2); and Estonia, Finland, Lithuania, Poland and Spain (Season 3)
Period: Overall Study
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Non-Influenza Comparator Vaccine
Started | 2258 | 2256
Completed | 2249 | 2247
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Non-Influenza Comparator Vaccine | Total
Number analyzed (Participants) | 2258 | 2256 | 4514
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (4.00) | 8.9 (4.11) | 8.8 (4.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1106 | 1082 | 2188
  Male | 1152 | 1174 | 2326
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 2245 | 2245 | 4490
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1106 | 1100 | 2206
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 1 | 0 | 1
  White | 1140 | 1139 | 2279
  More than one race | NA — Data field not captured in the eCRF | NA — Data field not captured in the eCRF | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 11 | 15 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Philippines | 902 | 898 | 1800
  Finland | 168 | 158 | 326
  Poland | 147 | 151 | 298
  Australia | 96 | 99 | 195
  Thailand | 201 | 199 | 400
  Lithuania | 142 | 150 | 292
  Estonia | 599 | 599 | 1198
  Spain | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy: First Occurrence of Either RT-PCR- or Culture-confirmed Influenza (Time-to-event Analyses) Due to Any Influenza Type A or B Strain Regardless of Antigenic Match to the Strains Selected for the Seasonal Vaccine in Subjects ≥2 to <18 Years
Description: The primary efficacy endpoint was defined as the time from the last study vaccination to the onset of the first occurrence of either RT-PCR- or culture-confirmed influenza (time-to-event analyses) due to any influenza Type A or B strain regardless of antigenic match to the strains selected for the seasonal vaccine, that occurred more than 14 days after the last vaccination until the end of the influenza season.
  Dataset Used: FAS-Efficacy = All subjects in the All Enrolled Set who received at least one dose of study vaccine and were evaluated for efficacy from 14 days after the last vaccination.
  The success criterion used for this primary objective was as follows: The efficacy of the QIVc was demonstrated if the lower limit (LL) of the 2-sided 95% confidence interval (CI) for VE was above 20%.
Time Frame: Day 14 to Day 180 or until the end of the influenza season, whichever is longer
Population: FAS Efficacy - All subjects in the All Enrolled Set who received at least one dose of study vaccine and were evaluated for efficacy from 14 days after the last vaccination.
Measure: Number; unit: Number of cases
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Non-Influenza Comparator Vaccine
Number analyzed (Participants) | 2257 | 2252
Number of cases | 175 | 364
Statistical Analysis 1: Comparison: QIVc (≥2 Years to <18 Years of Age) vs Non-Influenza Comparator Vaccine; Statistical Analysis title - Absolute Vaccine Efficacy Any Strain. Adjusted aVE for QIVc vs. comparator. Success criteria for the primary efficacy endpoint was met if the LL of the 2-sided 95% CI of the aVE estimate was greater than 20% (primary endpoint) using the protocol definition of ILI for the entire age range (2 to <18 years of age); Test type: Superiority — Success criterion were met as the LL of the 2-sided 95% CI was above 20%; Absolute Efficacy = 54.63, 95% CI 2-sided [45.67 to 62.12]

2. Primary Outcome: Co-Primary: First Occurrence of Either RT-PCR- or Culture-confirmed Influenza (Time-to-event Analyses) Due to Any Influenza Type A or B Strain Regardless of Antigenic Match to the Strains Selected for the Seasonal Vaccine in Subjects ≥3 to <18 Years
Description: The co-primary efficacy endpoint: was defined as the time from the last study vaccination to the onset of the first occurrence of either RT-PCR- or culture-confirmed influenza (time-to-event analyses) due to any influenza Type A or B strain regardless of antigenic match to the strains selected for the seasonal vaccine, that occurred more than 14 days after the last vaccination until the end of the influenza season.Absolute vaccine efficacy of QIVc by first occurrence RT-PCR or culture confirmed influenza, due to any influenza Type A and B strain in subjects ≥3 years to <18 years of age
Time Frame: Day 14 to Day 180 or until the end of the influenza season, whichever is longer
Population: as for outcome 1
Measure: Number; unit: Number of cases
Groups:
- QIVc (≥3 Years to <18 Years of Age): Cell-derived Seasonal Quadrivalent Influenza Vaccine
  QIVc: Cell-derived Quadrivalent Influenza Vaccine for intramuscular use containing each of the 2 influenza type A strains and each of the 2 influenza type B strains
Arm/Group | QIVc (≥3 Years to <18 Years of Age) | Non-Influenza Comparator Vaccine
Number analyzed (Participants) | 2208 | 2201
Number of cases | 171 | 351
Statistical Analysis 1: Comparison: QIVc (≥3 Years to <18 Years of Age) vs Non-Influenza Comparator Vaccine; Statistical analysis title - Absolute Vaccine Efficacy, Any Strain Adjusted aVE for QIVc vs. comparator. Success criteria for the primary efficacy endpoint was met if the LL of the 2-sided 95% CI of the aVE estimate was greater than 30% (co-primary endpoint) using the protocol definition of ILI for the entire age range (≥ 3 to <18 years of age); Test type: Superiority — Success criteria was met as the LL of the 2-sided 95% CI of the VE estimate was greater than 30% (co-primary endpoint); Absolute Vaccine Efficacy = 54.03, 95% CI 2-sided [44.8 to 61.71]

3. Secondary Outcome: Secondary Efficacy #1: First Occurrence of Either RT-PCR- or Culture-confirmed Influenza Due to Any Influenza Type A or B Strain Regardless of Antigenic Match to the Strains Selected for the Seasonal Vaccine
Description: The endpoint was defined as the time from the last study vaccination to the onset of the first occurrence of either RT-PCR- or culture-confirmed influenza due to any influenza Type A or B strain regardless of antigenic match to the strains selected for the seasonal vaccine, that occurred more than 14 days after the last vaccination until the end of the influenza season in subjects 2 to <18 years, 2 to <9 years, 4 to <18 years, and 9 to <18 years.
  Dataset used: FAS Efficacy = All subjects in the All Enrolled Set who received at least one dose of study vaccine and were evaluated for efficacy from 14 days after the last vaccination.
Time Frame: Day 14 to Day 180 or until the end of the influenza season, whichever is longer.
Population: FAS Efficacy = All subjects in the All Enrolled Set who received at least one dose of study vaccine and were evaluated for efficacy from 14 days after the last vaccination.
Measure: Number; unit: Number of cases
Groups:
- QIVc (≥2 Years to <9 Years of Age); QIVc (≥4 Years to <18 Years of Age); QIVc (≥9 Years to <18 Years of Age): Cell-derived Seasonal Quadrivalent Influenza Vaccine
  QIVc: Cell-derived Quadrivalent Influenza Vaccine for intramuscular use containing each of the 2 influenza type A strains and each of the 2 influenza type B strains
- Comparator (≥2 Years to <9 Years of Age); Comparator (≥4 Years to <18 Years of Age): Non-Influenza Comparator Vaccine
  Non-influenza Comparator Vaccine: Non-influenza comparator vaccine for intramuscular use
- Comparator (≥9 Years to <18 Years of Age): Non-influenza Comparator Vaccine:
  Non-influenza comparator vaccine for intramuscular use
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Non-Influenza Comparator Vaccine | QIVc (≥2 Years to <9 Years of Age) | Comparator (≥2 Years to <9 Years of Age) | QIVc (≥4 Years to <18 Years of Age) | Comparator (≥4 Years to <18 Years of Age) | QIVc (≥9 Years to <18 Years of Age) | Comparator (≥9 Years to <18 Years of Age)
Number analyzed (Participants) | 2257 | 2252 | 1146 | 1142 | 2045 | 2032 | 1111 | 1110
Number of cases | 175 | 364 | 123 | 234 | 154 | 310 | 52 | 130
Statistical Analysis 1: Comparison: QIVc (≥2 Years to <18 Years of Age) vs Non-Influenza Comparator Vaccine; Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 2 to <18yrs; Test type: Superiority — Statistical analysis description: Absolute Vaccine Efficacy (aVE) for 2 to <18 Years. Note that no prespecified criteria for success were defined for the secondary efficacy endpoints; Absolute Vaccine Efficacy = 54.63, 95% CI 2-sided [45.67 to 62.12]
Statistical Analysis 2: Comparison: QIVc (≥2 Years to <9 Years of Age) vs Comparator (≥2 Years to <9 Years of Age); Statistical analysis title: Absolute Vaccine Efficacy, Any Strain, 2 to <9yrs; Test type: Superiority — Statistical analysis description: Absolute Vaccine Efficacy (aVE) for 2 to <9 Years. Note that no prespecified criteria for success were defined for the secondary efficacy endpoints; Absolute Vaccine Efficacy = 50.51, 95% CI 2-sided [38.43 to 60.22]
Statistical Analysis 3: Comparison: QIVc (≥4 Years to <18 Years of Age) vs Comparator (≥4 Years to <18 Years of Age); Statistical analysis title: Absolute Vaccine Efficacy, Any Strain, 4 to <18yrs; Test type: Superiority — Statistical analysis description: Absolute Vaccine Efficacy (aVE) for 4 to <18 years. Note that no prespecified criteria for success were defined for the secondary efficacy endpoints; Absolute Vaccine Efficacy = 53.33, 95% CI 2-sided [43.38 to 61.54]
Statistical Analysis 4: Comparison: QIVc (≥9 Years to <18 Years of Age) vs Comparator (≥9 Years to <18 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 9 to <18yrs; Test type: Superiority — Statistical analysis description: Absolute Vaccine Efficacy (aVE) for 9 to <18 years. Note that no prespecified criteria for success were defined for the secondary efficacy endpoints; Absolute Vaccine Efficacy = 61.85, 95% CI 2-sided [47.37 to 72.34]

4. Secondary Outcome: Secondary Efficacy #2: First Occurrence of RT-PCR-confirmed Influenza Due to Any Influenza Type A or B Strain Regardless of Antigenic Match to the Strains Selected for the Seasonal Vaccine
Description: The endpoint was defined as the time from the last study vaccination to the onset of the first occurrence of RT-PCR-confirmed influenza due to any influenza Type A or B strain regardless of antigenic match to the strains selected for the seasonal vaccine, that occurred more than 14 days after the last vaccination until the end of the influenza season in subjects 2 to <18 years, 2 to <9 years, 4 to <18 years, and 9 to <18 years
  Dataset used: FAS Efficacy - All subjects in the All Enrolled Set who received at least one dose of study vaccine and were evaluated for efficacy from 14 days after the last vaccination.
Time Frame: Day 14 to Day 180 or until the end of the influenza season, whichever is longer.
Population: FAS-Efficacy = All subjects in the All Enrolled Set who received at least one dose of study vaccine and were evaluated for efficacy from 14 days after the last vaccination.
Measure: Number; unit: Number of cases
Groups:
- Comparator (≥9 Years to <18 Years of Age): Non-Influenza Comparator Vaccine
  Non-influenza Comparator Vaccine: Non-influenza comparator vaccine for intramuscular use
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Non-Influenza Comparator Vaccine | QIVc (≥2 Years to <9 Years of Age) | Comparator (≥2 Years to <9 Years of Age) | QIVc (≥4 Years to <18 Years of Age) | Comparator (≥4 Years to <18 Years of Age) | QIVc (≥9 Years to <18 Years of Age) | Comparator (≥9 Years to <18 Years of Age)
Number analyzed (Participants) | 2257 | 2252 | 1146 | 1142 | 2045 | 2032 | 1111 | 1110
Number of cases | 175 | 364 | 123 | 234 | 154 | 310 | 52 | 130
Statistical Analysis 1: Comparison: QIVc (≥2 Years to <18 Years of Age) vs Non-Influenza Comparator Vaccine; Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 2 to <18yrs; Test type: Superiority — Absolute Vaccine Efficacy (aVE) for 2 to <18 years. Note that no prespecified criteria for success were defined for the secondary efficacy endpoints; Absolute Vaccine Efficacy = 54.63, 95% CI 2-sided [45.67 to 62.12]
Statistical Analysis 2: Comparison: QIVc (≥2 Years to <9 Years of Age) vs Comparator (≥2 Years to <9 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 2 to <9yrs; Test type: Superiority — [test comment as in outcome 3, analysis 2]; Absolute Vaccine Efficacy = 60.78, 95% CI 2-sided [49.01 to 69.83]
Statistical Analysis 3: Comparison: QIVc (≥4 Years to <18 Years of Age) vs Comparator (≥4 Years to <18 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 4 to <18yrs; Test type: Superiority — [test comment as in outcome 3, analysis 3]; Absolute Vaccine Efficacy = 59.66, 95% CI 2-sided [49.08 to 68.05]
Statistical Analysis 4: Comparison: QIVc (≥9 Years to <18 Years of Age) vs Comparator (≥9 Years to <18 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 9 to <18yrs; Test type: Superiority — [test comment as in outcome 3, analysis 4]; Absolute Vaccine Efficacy = 60.72, 95% CI 2-sided [42.14 to 73.33]

5. Secondary Outcome: Secondary Efficacy #3: First Occurrence of Culture-confirmed Influenza Due to Any Influenza Type A or B Strain Regardless of Antigenic Match to the Strains Selected for the Seasonal Vaccine
Description: The secondary endpoint was defined as the time from the last study vaccination to the onset of the first occurrence of culture-confirmed influenza due to any influenza Type A or B strain regardless of antigenic match to the strains selected for the seasonal vaccine, that occurred more than 14 days after the last vaccination until the end of the influenza season in subjects 2 to <18 years, 2 to <9 years, 4 to <18 years, and 9 to <18 years.
  Dataset used: FAS Efficacy
Time Frame: Day 14 to Day 180 or until the end of the influenza season, whichever is longer.
Population: as for outcome 4
Measure: Number; unit: Number of cases
Groups:
- QIVc (≥2 Years to <9 Years of Age): Cell-derived Seasonal Quadrivalent Influenza Vaccine
  QIVc: Cell-derived Quadrivalent Influenza Vaccine for intramuscular use containing each of the 2 influenza type A strains and each of the 2 influenza type B strain
- QIVc (≥9 Years to <18 Years of Age): QIVc: Cell-derived Quadrivalent Influenza Vaccine
  for intramuscular use containing each of the 2 influenza type A strains and each of the 2 influenza type B strains
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Non-Influenza Comparator Vaccine | QIVc (≥2 Years to <9 Years of Age) | Comparator (≥2 Years to <9 Years of Age) | QIVc (≥4 Years to <18 Years of Age) | Comparator (≥4 Years to <18 Years of Age) | QIVc (≥9 Years to <18 Years of Age) | Comparator (≥9 Years to <18 Years of Age)
Number analyzed (Participants) | 2257 | 2252 | 1146 | 1142 | 2045 | 2032 | 1111 | 1110
Number of cases | 115 | 279 | 79 | 190 | 101 | 237 | 36 | 89
Statistical Analysis 1: Comparison: QIVc (≥2 Years to <18 Years of Age) vs Non-Influenza Comparator Vaccine; Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 2 to <18yrs; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Absolute Vaccine Efficacy = 60.81, 95% CI 2-sided [51.3 to 68.46]
Statistical Analysis 2: Comparison: QIVc (≥2 Years to <9 Years of Age) vs Comparator (≥2 Years to <9 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 2 to <9yrs; Test type: Superiority — [test comment as in outcome 3, analysis 2]; Absolute Vaccine Efficacy = 60.78, 95% CI 2-sided [49.01 to 69.83]
Statistical Analysis 3: Comparison: QIVc (≥4 Years to <18 Years of Age) vs Comparator (≥4 Years to <18 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 9 to <18yrs; Test type: Superiority — [test comment as in outcome 3, analysis 4]; Absolute Vaccine Efficacy = 59.66, 95% CI 2-sided [49.08 to 68.05]
Statistical Analysis 4: Comparison: QIVc (≥9 Years to <18 Years of Age) vs Comparator (≥9 Years to <18 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 9 to <18yrs; Test type: Superiority — [test comment as in outcome 3, analysis 4]; Absolute Vaccine Efficacy = 60.72, 95% CI 2-sided [42.14 to 73.33]

6. Secondary Outcome: Secondary Efficacy #4: First Occurrence of Culture-confirmed Influenza Due to Influenza Type A or B Strain Antigenically Matched to the Strains Selected for the Seasonal Vaccine
Description: The endpoint was defined as the time from the last study vaccination to the onset of the first occurrence of culture-confirmed influenza due to influenza Type A or B strain antigenically matched to the strains selected for the seasonal vaccine, that occurred more than 14 days after the last vaccination until the end of the influenza season in subjects 2 to <18 years, 2 to <9 years, 4 to <18 years, and 9 to <18 years.
Time Frame: Day 14 to Day 180 or until the end of the influenza season, whichever is longer.
Population: as for outcome 4
Measure: Number; unit: Number of cases
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Non-Influenza Comparator Vaccine | QIVc (≥2 Years to <9 Years of Age) | Comparator (≥2 Years to <9 Years of Age) | QIVc (≥4 Years to <18 Years of Age) | Comparator (≥4 Years to <18 Years of Age) | QIVc (≥9 Years to <18 Years of Age) | Comparator (≥9 Years to <18 Years of Age)
Number analyzed (Participants) | 2257 | 2252 | 1146 | 1142 | 2045 | 2032 | 1111 | 1110
Number of cases | 90 | 236 | 64 | 164 | 81 | 200 | 26 | 72
Statistical Analysis 1: Comparison: QIVc (≥2 Years to <18 Years of Age) vs Non-Influenza Comparator Vaccine; Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 2 to <18yrs; Test type: Superiority — [test comment as in outcome 3, analysis 1]; Absolute Vaccine Efficacy = 63.64, 95% CI 2-sided [53.64 to 71.48]
Statistical Analysis 2: Comparison: QIVc (≥2 Years to <9 Years of Age) vs Comparator (≥2 Years to <9 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 2 to <9yrs; Test type: Superiority — [test comment as in outcome 3, analysis 2]; Absolute Vaccine Efficacy = 63.04, 95% CI 2-sided [50.66 to 72.32]
Statistical Analysis 3: Comparison: QIVc (≥4 Years to <18 Years of Age) vs Comparator (≥4 Years to <18 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 4 to <18yrs; Test type: Superiority — [test comment as in outcome 3, analysis 3]; Absolute Vaccine Efficacy = 61.58, 95% CI 2-sided [50.25 to 70.53]
Statistical Analysis 4: Comparison: QIVc (≥9 Years to <18 Years of Age) vs Comparator (≥9 Years to <18 Years of Age); Statistical analysis title Absolute Vaccine Efficacy, Any Strain, 9 to <18yrs; Test type: Superiority — [test comment as in outcome 3, analysis 4]; Absolute Vaccine Efficacy = 64.78, 95% CI 2-sided [44.84 to 77.51]

7. Secondary Outcome: Secondary Immunogenicity: Geometric Mean Titers for 4 Influenza Strains (HI Assay)
Description: Immunogenicity was characterized by HI assay 3 weeks after the last vaccination in a subset of subjects 2 to <9 years of age enrolled in Season 2 (n=432) and Season 3 (n=319) who were immunized and had immunogenicity data at the assessed timepoints (FAS Immunogenicity). Immunogenicity was assessed at baseline (Day 1; all subjects in immunogenicity subset), at Day 22 (all "previously vaccinated" subjects receiving a single dose of the study vaccine), and at Days 29 and 50 (all "not previously vaccinated" subjects receiving 2 doses) for all 4 influenza strains using the HI assay.
Time Frame: Day 1 (all subjects), Day 22 (all previously vaccinated subjects) or Day 29 and Day 50 (all not previously vaccinated subjects receiving 2 doses)
Population: FAS Immunogenicity - All Subjects in the All Enrolled Set who received at least one dose of study vaccine and provided evaluable serum samples at both baseline at after the last vaccination
Measure: Number (95% Confidence Interval); unit: Geometric mean titers (GMTs)
Groups:
- QIVc (≥2 Years to <9 Years of Age) - Season 2; QIVc (≥2 Years to <9 Years of Age) - Season 3: Cell-derived Seasonal Quadrivalent Influenza Vaccine
  QIVc: Cell-derived Quadrivalent Influenza Vaccine for intramuscular use containing each of the 2 influenza type A strains and each of the 2 influenza type B strains
  ** Strain compositions recommended by the World Health Organization for the 2018-2019 Northern Hemisphere influenza season (WHO, 2018) for quadrivalent vaccines.
- Comparator (≥2 Years to <9 Years of Age) - Season 2; Comparator (≥2 Years to <9 Years of Age) - Season 3: Non-Influenza Comparator Vaccine
  Non-influenza Comparator Vaccine: Non-influenza comparator vaccine
Arm/Group | QIVc (≥2 Years to <9 Years of Age) - Season 2 | Comparator (≥2 Years to <9 Years of Age) - Season 2 | QIVc (≥2 Years to <9 Years of Age) - Season 3 | Comparator (≥2 Years to <9 Years of Age) - Season 3
Number analyzed (Participants) | 210 | 212 | 154 | 145
Geometric mean titers (GMTs)
  A/H1N1 Day 1 HI GMT | 50.83 [41.89 to 61.66] | 47.51 [39.15 to 57.64] | 36.62 [22.61 to 59.31] | 31.76 [19.88 to 50.74]
  A/H1N1 Day 22/50 HI GMT | 283.45 [249.22 to 322.38] | 49.20 [43.24 to 55.98] | 380.70 [283.12 to 511.91] | 48.22 [36.14 to 64.32]
  A/H3N2 Day 1 HI GMT | 97.02 [86.51 to 108.81] | 94.40 [84.19 to 105.84] | 20.85 [15.99 to 27.20] | 20.74 [16.02 to 26.85]
  A/H3N2 Day 22/50 HI GMT | 168.73 [150.87 to 188.70] | 96.27 [86.05 to 107.70] | 67.64 [57.03 to 80.24] | 16.73 [14.17 to 19.77]
  B/Victoria Day 1 HI GMT | 11.67 [9.97 to 13.67] | 11.73 [10.02 to 13.73] | 9.54 [7.25 to 12.54] | 9.41 [7.22 to 12.28]
  B/Victoria Day 22/50 HI GMT | 45.25 [39.73 to 51.54] | 11.94 [10.48 to 13.60] | 66.82 [51.29 to 87.04] | 11.94 [9.23 to 15.44]
  B/Yamagata Day 1 HI GMT | 10.87 [9.46 to 12.50] | 12.17 [10.59 to 13.99] | 23.98 [16.74 to 34.36] | 27.33 [19.27 to 38.76]
  B/Yamagata Day 22/50 HI GMT | 52.81 [45.77 to 60.94] | 12.34 [10.68 to 14.24] | 108.49 [85.16 to 138.22] | 21.68 [17.11 to 27.46]

8. Secondary Outcome: ISecondary Immunogenicity: Percentage of Subjects Achieving Seroconversion for 4 Influenza Strains (HI Assay)
Description: Immunogenicity was characterized by HI assay 3 weeks after the last vaccination in a subset of subjects 2 to <9 years of age enrolled in Season 2 (n=432) and Season 3 (n=319) who were immunized and had immunogenicity data at the assessed timepoints (FAS Immunogenicity). Immunogenicity was assessed at baseline (Day 1; all subjects in immunogenicity subset), at Day 22 (all "previously vaccinated" subjects receiving a single dose of the study vaccine), and at Days 29 and 50 (all "not previously vaccinated" subjects receiving 2 doses) for all 4 influenza strains using the HI assay.
  Seroconversion was defined as: either a prevaccination HI titer <1:10 and a postvaccination HI titer
  ≥1:40 or a prevaccination HI titer ≥1:10 and a ≥4 fold increase in postvaccination HI titer)
  Dataset used: FAS Immunogenicity = All subjects in the All Enrolled Set who received at least one dose of study vaccine and provided evaluable serum samples at both baseline and after the last vaccination.
Time Frame: Day 22 (all previously vaccinated subjects) or Day 29 and Day 50 (all not previously vaccinated subjects)
Population: FAS Immunogenicity: all subjects in the All Enrolled Set who received at least one dose of study vaccine and provided evaluable serum samples at both baseline and after the last vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Comparator (≥2 Years to <9 Years of Age): Non-Influenza Comparator Vaccine
  Non-influenza Comparator Vaccine: Non-influenza comparator vaccine
Arm/Group | QIVc (≥2 Years to <9 Years of Age) - Season 2 | Comparator (≥2 Years to <9 Years of Age) | QIVc (≥2 Years to <9 Years of Age) - Season 3 | Non-Influenza Comparator Vaccine
Number analyzed (Participants) | 210 | 212 | 154 | 145
Percentage of participants
  A/H1N1 | 59.5 [52.55 to 66.22] | 1.9 [0.52 to 4.80] | 74.0 [66.35 to 80.75] | 6.2 [2.88 to 11.46]
  A/H3N2 | 19.0 [13.97 to 25.02] | 1.9 [0.52 to 4.80] | 51.9 [43.76 to 60.06] | 1.4 [0.17 to 4.89]
  B/Victoria | 40.0 [33.32 to 46.97] | 2.9 [1.06 to 6.11] | 58.4 [50.23 to 66.32] | 3.4 [1.13 to 7.86]
  B/Yamagata | 49.5 [42.57 to 56.49] | 4.8 [2.31 to 8.58] | 58.4 [50.23 to 66.32] | 1.4 [0.17 to 4.89]

9. Secondary Outcome: Secondary Immunogenicity: Geometric Mean Ratio for 4 Influenza Strains (HI Assay)
Description: Immunogenicity was characterized by HI assay 3 weeks after the last vaccination in a subset of subjects 2 to <9 years of age enrolled in Season 2 (n=432) and Season 3 (n=319) who were immunized and had immunogenicity data at the assessed timepoints (FAS Immunogenicity). Immunogenicity was assessed at baseline (Day 1; all subjects in immunogenicity subset), at Day 22 (all "previously vaccinated" subjects receiving a single dose of the study vaccine), and at Days 29 and 50 (all "not previously vaccinated" subjects receiving 2 doses) for all 4 influenza strains using the HI assay.
  Geometric mean ratios (GMRs) measure the ratio in immunogenicity titers within subject\
  Dataset used: FAS Immunogenicity = All subjects in the All Enrolled Set who received at least one dose of study vaccine and provided evaluable serum samples at both baseline and after the last vaccination.
Time Frame: Day 22/Day 1 (all previously vaccinated subjects) or Day 29/Day 1 and Day 50/Day 1 (all not previously vaccinated subjects receiving 2 doses)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Geometric mean ratio (GMR)
Groups:
- QIVc (≥2 Years to <9 Years of Age) - Season 2: Cell-derived Seasonal Quadrivalent Influenza Vaccine
  QIVc: Cell-derived Quadrivalent Influenza Vaccine for intramuscular use containing each of the 2 influenza type A strains and each of the 2 influenza type B strains
Arm/Group | QIVc (≥2 Years to <9 Years of Age) - Season 2 | Comparator (≥2 Years to <9 Years of Age) - Season 2 | QIVc (≥2 Years to <9 Years of Age) - Season 3 | Comparator (≥2 Years to <9 Years of Age) - Season 3
Number analyzed (Participants) | 210 | 212 | 154 | 145
Geometric mean ratio (GMR)
  A/H1N1 | 5.76 [5.06 to 6.55] | 1.00 [0.88 to 1.14] | 9.73 [7.24 to 13.09] | 1.23 [0.92 to 1.64]
  A/H3N2 | 1.74 [1.56 to 1.95] | 0.99 [0.89 to 1.11] | 4.14 [3.49 to 4.91] | 1.02 [0.87 to 1.21]
  B/Victoria | 3.79 [3.33 to 4.32] | 1.00 [0.88 to 1.14] | 7.01 [5.38 to 9.14] | 1.25 [0.97 to 1.62]
  B/Yamagata | 4.63 [4.01 to 5.34] | 1.08 [0.94 to 1.25] | 5.27 [4.14 to 6.72] | 1.05 [0.83 to 1.33]

10. Secondary Outcome: Secondary Immunogenicity: Percentage of Subjects With HI Titer ≥1:40 for All 4 Influenza Strains (HI Assay)
Description: Immunogenicity was characterized by HI assay 3 weeks after the last vaccination in a subset of subjects 2 to <9 years of age enrolled in Season 2 (n=432) and Season 3 (n=319) who were immunized and had immunogenicity data at the assessed timepoints (FAS Immunogenicity). Immunogenicity was assessed at baseline (Day 1; all subjects in immunogenicity subset), at Day 22 (all "previously vaccinated" subjects receiving a single dose of the study vaccine), and at Days 29 and 50 (all "not previously vaccinated" subjects receiving 2 doses) for all 4 influenza strains using the HI assay.
  The measures for assessing immunogenicity as determined by HI were as follows: Percentage of subjects with an HI titer ≥1:40 on Day 22 (all "previously vaccinated" subjects receiving a single vaccine dose) or Days 29 and 50 (all "not previously vaccinated" subjects receiving 2 doses) for all 4 influenza strains
Time Frame: Day 1 (all subjects), Day 22 (all "previously vaccinated" subjects receiving a single vaccine dose) or Days 29 and 50 (all "not previously vaccinated"subjects receiving 2 doses)
Population: Dataset used: FAS Immunogenicity = all subjects in the All Enrolled Set who received at least one dose of study vaccine and provided evaluable serum samples at both baseline and after the last vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | QIVc (≥2 Years to <9 Years of Age) - Season 2 | Comparator (≥2 Years to <9 Years of Age) - Season 2 | QIVc (≥2 Years to <9 Years of Age) - Season 3 | Comparator (≥2 Years to <9 Years of Age) - Season 3
Number analyzed (Participants) | 210 | 212 | 154 | 145
Percentage of participants
  A/H1N1 | 88.6 [83.47 to 92.54] | 58.6 [51.59 to 65.31] | 94.8 [90.02 to 97.73] | 55.2 [46.70 to 63.43]
  A/H3N2 | 90.0 [85.12 to 93.70] | 92.4 [87.92 to 95.58] | 74.0 [66.35 to 80.75] | 24.8 [18.03 to 32.68]
  B/Victoria | 54.3 [47.29 to 61.16] | 24.30 [18.65 to 30.66] | 68.8 [60.88 to 76.04] | 13.1 [8.08 to 19.70]
  B/Yamagata | 63.8 [56.91 to 70.31] | 21.4 [16.08 to 27.60] | 79.2 [71.95 to 85.33] | 46.2 [37.90 to 54.67]

11. Secondary Outcome: Safety: Percentage of Subjects With Solicited Local and Systemic Adverse Events for 7 Days After Vaccination
Description: The measures for assessing safety and tolerability were as follows: Percentage of subjects with solicited local and systemic adverse events (AEs) for 7 days after vaccination on Day 1 (for "previously vaccinated" subjects) or for 7 days after vaccination on Day 1 and Day 29 (for "not previously vaccinated" subjects) in the QIVc group and the non-influenza comparator vaccine group.
  Dataset used: Solicited Safety Set
Time Frame: days after vaccination on Day 1 (for "previously vaccinated" subjects) or for 7 days after vaccination on Day 1 and Day 29 (for "not previously vaccinated" subjects)
Population: Dataset used: Solicited Safety Set = All subjects in the Exposed Set who had gone through any assessment of local and systemic site reaction and/or assessment of any use of analgesics/antipyretics.
  Note: Other solicited adverse events refer to use of analgesics / antipyretics for prophylaxis or treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Comparator (≥2 Years to <18 Years of Age): Non-Influenza Comparator Vaccine
  Non-influenza Comparator Vaccine: Non-influenza comparator vaccine
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Comparator (≥2 Years to <18 Years of Age)
Number analyzed (Participants) | 2255 | 2254
Percentage of participants
  Solicited AEs | 51.4 | 48.6
  Solicited Local AEs | 36.8 | 33.6
  Solicited Systemic AEs | 31.4 | 30.5
  Other | 8.6 | 7.3

12. Secondary Outcome: Safety: Percentage of Subjects With Unsolicited AEs for 21 Days After Vaccination
Description: The measures for assessing safety and tolerability were as follows: Percentage of subjects with unsolicited AEs assessed from Day 1 to Day 22 (for "previously vaccinated" subjects) or from Day 1 to Day 50 (for "not previously vaccinated" subjects) in the QIVc group and the non-influenza comparator vaccine group.
  Dataset used: Unsolicited Safety Set (Unsolicited Adverse Events)
Time Frame: Day 1 to Day 22 (for previously vaccinated subjects) or Day 1 to Day 50 (for not previously vaccinated subjects)
Population: Dataset used: unsolicited Safety Set defined as all subjects in the Exposed Set who had gone through any AE assessments, ie, a subject did not have to have any AEs to be included in this population
Measure: Number; unit: Percentage of participants
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Comparator (≥2 Years to <18 Years of Age)
Number analyzed (Participants) | 2258 | 2255
Percentage of participants
  Any AE | 28.0 | 27.9
  Any AE (Mild) | 24.4 | 24.6
  Any AE (Moderate) | 4.8 | 4.5
  Any AE (Severe) | 0.5 | 0.5
  Related AE | 4.3 | 3.9

13. Secondary Outcome: Safety: Subjects With SAEs, AEs Leading to Withdrawal From Vaccination and/or the Study,(MAAEs) Within 30 Days of a 1st Occurrence, Post-ILI, and NOCDs Reported During Entire Study Participation or End of Flue Season, Whichever Was Longer
Description: The measures for assessing safety and tolerability were as follows: Percentage of subjects with SAEs, AEs leading to withdrawal from vaccination and/or the study, Medically-Attended AEs (MAAEs) within 30 days after the first occurrence of an ILI, and New Onset of Chronic Diseases (NOCDs) reported during the subject's entire participation in the study (ie, from Day 1 to Day 181 [for "previously vaccinated" subjects] or from Day 1 to Day 209 [for "not previously vaccinated" subjects]), or until the end of influenza season, whichever was longer, and all medications associated with these events.
  Dataset used: Overall Safety Set
Time Frame: Day 1 to Day 181 (for previously vaccinated subjects) or to Day 209 (for not previously vaccinated subjects)
Population: Dataset used: overall safety set defined as all subjects in the Solicited Safety Set and/or Unsolicited Safety Set. Subjects providing only 30 minutes postvaccination safety data were also reported separately in a 30-minute postvaccination safety analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Comparator (≥2 Years to <18 Years of Age)
Number analyzed (Participants) | 2258 | 2255
Percentage of participants
  SAE | 1.1 | 1.3
  Related SAE | 0 | 0
  AE leading to study withdrawal | 0 | 0
  MAAE | 27.2 | 30.1
  NOCD | 0.4 | 0.5
  Death | 0 | 0.04

ADVERSE EVENTS:
Time Frame: Day 1 through end of study
Description: Adverse event reporting additional description: Nonserious Unsolicited AEs and SAEs are reported
Arm/Group | QIVc (≥2 Years to <18 Years of Age) | Non-Influenza Comparator Vaccine
All-Cause Mortality (participants affected / at risk) | 0/2258 | 1/2255
Serious Adverse Events (participants affected / at risk) | 25/2258 | 30/2255
Other Adverse Events (participants affected / at risk) | 871/2258 | 963/2255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QIVc (≥2 Years to <18 Years of Age) (N=2258) | Non-Influenza Comparator Vaccine (N=2255)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neuropathy, peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 0 (0)
Brain Edema (Nervous system disorders) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Status Migrainosus (Nervous system disorders) | 0 (0) | 1 (1)
Unevaluable event (General disorders) | 1 (1) | 0 (0)
Anorexia nervosa (Psychiatric disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type I Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Chronic Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Dengue fever (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia mycoplasma (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Dengue hemorrhagic fever (Infections and infestations) | 1 (1) | 1 (1)
Enterococcal Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QIVc (≥2 Years to <18 Years of Age) (N=2258) | Non-Influenza Comparator Vaccine (N=2255)
Influenza like illness (General disorders) | 791 (791) | 894 (894)
Nasopharyngitis (Infections and infestations) | 111 (111) | 135 (135)
Upper respiratory tract infection (Infections and infestations) | 298 (298) | 270 (270)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03165617/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT03165617/SAP_001.pdf